CLINICAL TRIAL: NCT00386022
Title: The Effect of Aging on the Isolated Pituitary Response to Gonadotropin Releasing Hormone at Baseline and With Low Dose Estrogen Administration
Brief Title: The Effects of Aging and Estrogen on the Pituitary
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Associate Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2000-P-002498; R01AG013241 (NIH)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Gonadotropin-releasing hormone; Estrogens; postmenopausal women; Pituitary hormones
MeSH Terms: interventions — Gonadotropin-Releasing Hormone; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Estradiol

STUDY DESIGN:
Intervention Model Description: The study will is considered sequential as participants were studied at baseline and after one month of low-dose estrogen. Randomization refers to randomization of the order of doses of GnRH between participants.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young postmenopausal women (Experimental): intervention: graded doses of GnRH following NAL-GLU GnRH antagonist administration with or without transdermal estrogen patch
  Interventions: Drug: GnRH; Drug: NAL-GLU GnRH antagonist; Drug: Estrogen patch
- Older postmenopausal women (Experimental): intervention: graded doses of GnRH following NAL-GLU GnRH antagonist administration with or without transdermal estrogen patch
  Interventions: Drug: GnRH; Drug: NAL-GLU GnRH antagonist; Drug: Estrogen patch

INTERVENTIONS:
Drug: GnRH — GnRH doses of 25, 75, 250 and 750 ng/kg will be given IV every 4 hr at baseline and after transdermal estradiol
  Other Names: gonadotropin-releasing hormone; Factryl
Drug: NAL-GLU GnRH antagonist — A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg before and after transdermal estradiol
  Other Names: GnRH antagonist
Drug: Estrogen patch — transdermal estrogen patches 0.05mg/day, changing the patch every 86 hr in second part of sequential study
  Other Names: Climara; Estraderm

SUMMARY:
The purpose of this study is to study the effects of aging and estrogen on the brain. Specifically, this study will examine how the hypothalamus signals the pituitary gland to secrete reproductive hormones and how that changes with aging.

DETAILED DESCRIPTION:
Although it is clear that loss of ovarian function plays a major role in the menopause in women, there is evidence from animal studies that primary age-related hypothalamic and pituitary changes may also contribute to reproductive aging. Complete cessation of ovarian function results in the loss of negative feedback of ovarian steroids and inhibin on the hypothalamic and pituitary components of the reproductive axis. An increase in serum levels of luteinizing hormone (LH) and follicle-stimulating hormone (FSH) occurs in postmenopausal women with removal of negative ovarian feedback. However, levels of LH and FSH after menopause decline steadily as a function of age in most though not all studies.

The current study is designed to determine: 1) whether negative feedback on LH and FSH occurs at the pituitary; and 2) whether there is an effect of aging on estrogen negative feedback at the pituitary. Younger and older postmenopausal women underwent a baseline study and a second identical study after a month of low dose estrogen replacement. The study protocol consisted of the following: 1) administration of a GnRH antagonist (Nal-Glu at 150 mg/kg that blocks endogenous GnRH so that the dose and interval of pituitary exposure to GnRH are precisely controlled; 2) beginning 8 hours following GnRH antagonist administration (at a time when LH had reached its nadir following GnRH receptor blockade), administration of 4 graded doses of GnRH (25, 75, 250 and 750 ng/kg every 2 hours with 2 hours of blood draws following each dose). Blood was sampled every 30 min for 4 hours before antagonist administration, every 30 min for the following 7 hours and then every 10 min until the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* 45-55 or 70-80 years old
* History of natural menopause defined by the absence of menses for at least 12 months (or history of surgical menopause defined as bilateral oophorectomy) and a FSH level >26 IU/L
* On no hormonal medication or herbal supplements and/or over the counter menopause therapy for a minimum of 2 months prior to study
* Normal thyroid stimulating hormone, prolactin, factor V Leiden, and complete blood count - Normal blood urea nitrogen and creatinine (< 2 times the upper limit of normal)
* basal metabolic index ≤ 30
* Non-smokers or smoke less than 10 cigarettes/day

Exclusion Criteria:

* Absolute contraindications to the use of physiologic replacement doses of estrogen, including a negative screening mammogram within the past 24 months
* History of coronary artery disease
* On medications thought to act centrally on the GnRH pulse generator
* Past history of hypersensitivity or allergy to narcotics, vancomycin, muscle relaxants, aspirin, and/or anaphylactic reaction(s) to other drugs
* Prior history of breast cancer and/or blood clots

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-01; Primary Completion 2012-01 (Actual); Study Completion 2018-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded data with identifying information can be requested by contacting the PI.

REFERENCES:
- [Result] Shaw ND, Histed SN, Srouji SS, Yang J, Lee H, Hall JE. Estrogen negative feedback on gonadotropin secretion: evidence for a direct pituitary effect in women. J Clin Endocrinol Metab. 2010 Apr;95(4):1955-61. doi: 10.1210/jc.2009-2108. Epub 2010 Feb 4. PMID 20133465
- [Result] Shaw ND, Srouji SS, Histed SN, McCurnin KE, Hall JE. Aging attenuates the pituitary response to gonadotropin-releasing hormone. J Clin Endocrinol Metab. 2009 Sep;94(9):3259-64. doi: 10.1210/jc.2009-0526. Epub 2009 Jun 23. PMID 19549740

RESULTS

PARTICIPANT FLOW:
Groups:
- Younger PMW: Postmenopausal women (PMW) 45-55 years old receiving the following series of treatments:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
  Participants studied at baseline (period 1) and after 1 month of transdermal estrogen 0.05 mg/day (period 2)
- Older PMW: Postmenopausal women (PMW) 70-80 years old receiving the following series of treatments:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
  Participants studied at baseline (period 1) and after 1 month of transdermal estrogen 0.05 mg/day (period 2)
Period: Baseline
Arm/Group | Younger PMW | Older PMW
Started | 10 | 9
All Doses of GnRH | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Plus Estrogen
Arm/Group | Younger PMW | Older PMW
Started | 10 | 9
Estrogen Patch | 8 | 9
All Doses GnRH | 8 | 8
Completed | 8 | 8
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Healthy postmenopausal women who experienced their last menstrual period a minimum of 12 months previously and met all inclusion and exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Younger PMW | Older PMW | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (2.46) | 72.8 (2.88) | 61.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pituitary Response to GnRH
Description: Baseline LH and FSH responses to each of 4 GnRH doses - peak to nadir amplitude expressed as percent (%) change from nadir
Time Frame: Peak hormone level within 2 hours post GnRH doses
Measure: Mean (Standard Error); unit: Percent change
Groups:
- Younger PMW: Postmenopausal women aged 45-55 years studied at baseline using the following interventions:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
- Older PMW: Postmenopausal women aged 70-80 years studied at baseline using the following interventions:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
Arm/Group | Younger PMW | Older PMW
Number analyzed (Participants) | 10 | 9
Percent change
  LH % change: 25 ng/kg GnRH | 7.88 (1.76) | 6.00 (1.49)
  LH % change: 75 ng/kg GnRH | 20.08 (2.94) | 17.27 (3.65)
  LH % change: 250 ng/kg GnRH | 62.82 (12.15) | 43.96 (5.70)
  LH % change: 750 ng/kg GnRH | 137.51 (14.17) | 103.73 (8.60)
  FSH % change 25 ng/kg GnRH | 5.30 (.88) | 4.32 (.89)
  FSH % change: 75 ng/kg GnRH | 8.01 (1.13) | 6.98 (1.26)
  FSH % change: 250 ng/kg GnRH | 14.57 (1.87) | 9.29 (1.32)
  FSH % change: 750 ng/kg | 23.55 (1.82) | 17.53 (2.40)
Statistical Analysis 1: Comparison: Younger PMW vs Older PMW; Test type: Equivalence — null hypothesis will be accepted if there is no difference in the LH response to GnRH as a function of dose in young or old postmenopausal women; p < 0.001, Repeated measures ANCOVA — LH % change with dose
Statistical Analysis 2: Comparison: Younger PMW vs Older PMW; null hypothesis: there will be no difference in the LH and FSH responses to graded doses of GnRH between younger and older postmenopausal women; Test type: Equivalence — null hypothesis will be accepted if there is no difference in the LH response to GnRH between younger and older postmenopausal women; p < 0.03, Repeated measures ANCOVA — LH % change with age
Statistical Analysis 3: Comparison: Younger PMW vs Older PMW; Test type: Equivalence — null hypothesis will be accepted if there is no difference in the FSH response to GnRH as a function of dose in younger or older postmenopausal women; p < 0.001, Repeated measures ANCOVA — FSH % change with dose
Statistical Analysis 4: Comparison: Younger PMW vs Older PMW; Test type: Equivalence — null hypothesis will be accepted if there is no difference in the FSH response to GnRH between young and old postmenopausal women; p < 0.005, Repeated measures ANCOVA — FSH % change with age

2. Primary Outcome: Effect of Estrogen on Pituitary Response to GnRH
Description: LH and FSH responses to each of 4 GnRH doses, expressed as change in amplitude [amp] from peak to nadir between plus estrogen and baseline conditions
Time Frame: Peak hormone level within 2 hours post GnRH doses
Measure: Mean (Standard Error); unit: IU/L
Groups:
- Young Postmenopausal Women: Postmenopausal women aged 45-55 years studied after 1 month of transdermal estrogen 0.05 mg/day using the following interventions:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
- Older Postmenopausal Women: Postmenopausal women aged 70-80 years studied after 1 month of transdermal estrogen 0.05 mg/day using the following interventions:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
Arm/Group | Young Postmenopausal Women | Older Postmenopausal Women
Number analyzed (Participants) | 8 | 8
IU/L
  LH amp change: 25 ng/kg GnRH | -0.38 (1.9) | -0.53 (1.0)
  LH amp change: 75 ng/kg GnRH | -2.9 (3.1) | -0.54 (1.7)
  LH amp change: 250 ng/kg GnRH | -17.8 (8.0) | -5.4 (3.4)
  LH amp change: 750 ng/kg GnRH | -27.1 (18.8) | -14.2 (4.6)
  FSH amp change: 25 ng/kg GnRH | -2.7 (1.9) | -0.6 (1.3)
  FSH amp change: 75 ng/kg | -6.7 (7.5) | 0.21 (1.8)
  FSH amp change: 250 ng/kg | -12.1 (3.3) | -1.9 (2.2)
  FSH amp change: 750 ng/kg | -15.4 (3.9) | -5.8 (3.3)
Statistical Analysis 1: Comparison: Young Postmenopausal Women vs Older Postmenopausal Women; Test type: Equivalence — null hypothesis will be accepted if there is no effect of estrogen on the LH response to GnRH in younger and older postmenopausal women; p < 0.01, Repeated measured ANCOVA — LH amplitude response with estrogen
Statistical Analysis 2: Comparison: Young Postmenopausal Women vs Older Postmenopausal Women; Test type: Equivalence — The null hypothesis will be accepted if there is no effect of estrogen on the FSH response to GnRH in younger and older postmenopausal women; p < 0.0001, Repeated measures ANCOVA — FSH amplitude response with estrogen
Statistical Analysis 3: Comparison: Young Postmenopausal Women vs Older Postmenopausal Women; Test type: Equivalence — The null hypothesis will be accepted if there is no effect of age on the effect of estrogen on the FSH response to GnRH; p < 0.02, Repeated measures ANCOVA — FSH amplitude response to estrogen with age
Statistical Analysis 4: Comparison: Young Postmenopausal Women vs Older Postmenopausal Women; Test type: Equivalence — The null hypothesis will be accepted if there is no effect of age on the effect of estrogen on the LH response to GnRH; p = 0.4, Repeated measures ANCOVA — LH amplitude response to estrogen with age

ADVERSE EVENTS:
Time Frame: 3 months
Description: Information on AEs was collected for a 3 month period from study entry for each subject.
Groups:
- Younger PMW: Postmenopausal women aged 45-55 years studied at baseline (period 1) and after 1 month of transdermal estrogen 0.05 mg/day (period 2) using the following interventions:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
- Older PMW: Postmenopausal women aged 70-80 years studied at baseline (period 1) and after 1 month of transdermal estrogen 0.05 mg/day (period 2) using the following interventions:
  1. A single subcutaneous injection of the NAL-GLU GnRH antagonist at a dose of 150 mcg/kg.
  2. GnRH doses of 25, 75, 250 and 750 ng/kg given IV every 4 hr
Arm/Group | Younger PMW | Older PMW
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/9
Other Adverse Events (participants affected / at risk) | 2/10 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger PMW (N=10) | Older PMW (N=9)
New Onset Rapid Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — On admission to Visit #2, subject's heart rate was 155 bpm. EKG revealed subject was in new onset rapid atrial fibrillation. Subject denied symptoms; transferred to a telemetry floor for rate control and discharged 2 days later. PCP notified.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger PMW (N=10) | Older PMW (N=9)
fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient slipped on ice and twisted knee
genital herpes diagnosis (Infections and infestations) | 1 (1) | 0 (0) — diagnosis of genital herpes after baseline visit

LIMITATIONS AND CAVEATS:
No significant limitations were present in this study and the subsequent analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No